CLINICAL TRIAL: NCT04343326
Title: The Additional Role of Supplemental Oxygen Therapy in Accelerated Corneal Collagen Cross-linking in Progressive Keratoconus. A Randomized Clinical Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of department, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 9900
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- accelerated corneal cross linking+ delivery of systemic oxygen (Active Comparator): corneal cross linking is performed using an accelerated protocol (9 mW/ CM2 for 10 minutes) in addition to the delivery of systemic oxygen with a rate of 5 liters/min through a nasal mask for 10 minutes during UV-A ablation
  Interventions: Procedure: perform corneal collagen cross linking accelerated and delivery of systemic oxygen
- accelerated corneal collagen cross-linking (Active Comparator): corneal cross linking with the same accelerated protocol without additional oxygen therapy.
  Interventions: Procedure: perform corneal collagen cross linking accelerated and without additional oxygen therapy
- conventional corneal collagen cross-linking (Active Comparator): Conventional corneal cross linking using 30 mW/CM2 UV-A ablation for 30 minutes
  Interventions: Procedure: perform Conventiona corneal collagen cross linking

INTERVENTIONS:
Procedure: perform corneal collagen cross linking accelerated and delivery of systemic oxygen — CXL is performed using an accelerated protocol (9 mW/ CM2 for 10 minutes) in addition to the delivery of systemic oxygen with a rate of 5 liters/min through a nasal mask for 10 minutes during UV-A ablation
  Arms: accelerated corneal cross linking+ delivery of systemic oxygen
Procedure: perform corneal collagen cross linking accelerated and without additional oxygen therapy — corneal collagen cross linking with accelerated protocol without additional oxygen therapy
  Arms: accelerated corneal collagen cross-linking
Procedure: perform Conventiona corneal collagen cross linking — Conventional CXL using 30 mW/CM2 UV-A ablation for 30 minutes
  Arms: conventional corneal collagen cross-linking

SUMMARY:
It is aimed to investigate the role of supplemental systemic oxygen therapy during accelerated corneal collagen crosslinking (CXL).

In this prospective randomized clinical trial, patients with progressive keratoconus who are candidates for receiving CXL will be included. The patients will be randomized and allocated to three different CXL protocol. In the first group (OA-CXL), CXL is performed using an accelerated protocol (9 mW/ CM2 for 10 minutes) in addition to the delivery of systemic oxygen with a rate of 5 liters/min through a nasal mask for 10 minutes during UV-A ablation. Patients in the second group (A-CXL) will receive CXL with the same accelerated protocol without additional oxygen therapy. Conventional CXL using 30 mW/CM2 UV-A ablation for 30 minutes is perfomed in the patients of the third goup (C-CXL). Maximum keratometry in Sirius corneal tomography as the primary outcome and uncorrected and corrected distance visual acuity (UDVA, CDVA) and corneal biomechanical properties including corneal resistance factor (CRF) and corneal hysteresis (CH) as secondary outcome measures are followed for a six- and 12-months period. A P-value of less than 0.05 is considered as statistically significance level.

ELIGIBILITY:
Inclusion Criteria:

* definitive diagnosis of progressive keratoconus for whom CXL is indicated were enrolled in this study
* The indication is identified by a cornea specialist and was considered as follows.
* Patients with the definitive diagnosis of KC who aged 18 or more were considered for the procedure if they had an increase of 1 D in Kmax or an increase of 1D in the manifest cylinder over the past 12 months.

Exclusion Criteria:

* patients with the previous history of corneal surgery
* corneal scar or pathologies like herpetic eye disease or severe dry eye
* corneal thickness less than 400 micrometers
* pregnant or nursing women
* corneal Kmax more than 60
* age over 35 years
* severe ocular surface disease

Max Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative refractive error | 12 months
  Sirius and ocular response analyzer

SECONDARY OUTCOMES:
Ocular biomechanics | 6 months
  Ocular response analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Faramarzi A, Hassanpour K, Rahmani B, Yazdani S, Kheiri B, Sadoughi MM. Systemic supplemental oxygen therapy during accelerated corneal crosslinking for progressive keratoconus: randomized clinical trial. J Cataract Refract Surg. 2021 Jun 1;47(6):773-779. doi: 10.1097/j.jcrs.0000000000000513. PMID 33252568